CLINICAL TRIAL: NCT02087280
Title: Metabolic Phenotyping to Predict Risk of Relapse in Patients With Anorexia Nervosa
Brief Title: Metabolic Phenotyping in Anorexia Nervosa
Status: Withdrawn | Type: Observational
Why Stopped: We did not receive funding
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Forschungegemeinschaft (Unknown)
Responsible Party: Principal Investigator, Dr. Verena Haas, Dr. oec. troph. Verena Haas, Charite University, Berlin, Germany
Other Study IDs: VHaas; HA 7034/2-1 (Other: Deutsche Forschungsgemeinschaft)
Record Dates: First submitted 2014-01-03; First posted 2014-03-14 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarkers of energy metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anorexia Nervosa
- Healthy controls

SUMMARY:
After discharge from inpatient treatment, 30-50% of patients with Anorexia Nervosa require re-hospitalization within 4-12 months. So far, high relapse rates are mostly considered as lack of the patient's compliance and motivation to recover. However in studies, psychological relapse predictors explain only a minor part of the variance in relapse risk. Metabolic phenotyping has clinical value to predict weight course in obese patients and we assume that it could also be clinically relevant in patients with AN. We hypothesize that in patients with a dissipative but not with the thrifty phenotype, positive energy balance during refeeding causes an over proportional rise in energy expenditure, counteracts continuous weight gain during inpatient treatment, and increases relapse risk within one year after discharge. Thus we believe that metabolic phenotype as a biological parameter has prognostic value for the disease course in AN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Anorexia Nervosa
* Between 12 and 18 years of age
* Written and informed consent of patient and parents
* Mental ability to understand the concept of the study
* Inpatient admission to Charité University Clinic with body weight below the 10th BMI-Percentile

Exclusion Criteria:

* Any further disease other than AN with significant influence on body composition and energy metabolism or its assessment

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female adolescents with Anorexia Nervosa
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Relapse | 1 year after discharge

SECONDARY OUTCOMES:
Metabolic phenotype | Baseline (during inpatient stay)
Biomarkers | Baseline (during inpatient stay)

CONTACTS AND LOCATIONS:
Overall Officials: Verena K Haas, PhD, Principal Investigator — Charité University Berlin
Locations (1):
- Charité University Clinic, Berlin, Germany

REFERENCES:
- [Derived] Haas V, Stengel A, Mahler A, Gerlach G, Lehmann C, Boschmann M, de Zwaan M, Herpertz S. Metabolic Barriers to Weight Gain in Patients With Anorexia Nervosa: A Young Adult Case Report. Front Psychiatry. 2018 May 18;9:199. doi: 10.3389/fpsyt.2018.00199. eCollection 2018. PMID 29867616